CLINICAL TRIAL: NCT05255627
Title: The Effect Of The Mobıle Applıcatıon On Nursıng Students On Preventıon, Treatment And Care Of Pressure Injury
Brief Title: Mobile Application Effectiveness in Pressure Injury Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, PhD RN Assistant Professor Hamiyet KIZIL, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15032021
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Knowledge; Satisfaction
Keywords: knowledge; Satisfaction; pressure injury
MeSH Terms: conditions — Personal Satisfaction; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): "Prevention, Care and Treatment of Pressure Injury" was explained by 1 researcher who is responsible for the Nursing Fundamentals course, using written educational material prepared in line with the literature.
  Interventions: Other: Control
- Mobile application group (Experimental Group) (Experimental): A mobile application program was installed on their phones for the experimental group students to benefit from. "Prevention, Care and Treatment of Pressure Injury" was explained by 1 researcher who is responsible for the Nursing Fundamentals course, using a mobile application program prepared in line with the literature.
  Interventions: Other: Mobile application group (Experimental Group)

INTERVENTIONS:
Other: Control — "Prevention, Care and Treatment of Pressure Injury" was explained by 1 researcher who is responsible for the Nursing Fundamentals course, using written educational material prepared in line with the literature.
  Arms: Control Group
Other: Mobile application group (Experimental Group) — A mobile application program was installed on the phones of the experimental group students for their benefit. "Prevention, Care and Treatment of Pressure Injury" was explained by 1 researcher who is responsible for the Nursing Fundamentals course, using a mobile application program prepared in line with the literature.
  Arms: Mobile application group (Experimental Group)

SUMMARY:
The research was designed in a randomized controlled experimental type in order to determine the effect of mobile application on students' knowledge levels and satisfaction levels about the prevention, treatment and care of pressure injuries. The population of the study conducted in the fall semester of the 2020-2021 academic year consisted of students enrolled in the Basic Principles and Practices in Nursing course at a foundation university in Istanbul between March and June 2021 (N=78). The sample size was calculated with G power 3.1.9.4, based on similar studies, and it was calculated that at least 28 people should be included in each group, with the pre-acceptance of α error being 5%, research power (power) 80%, and an effect value of 0.77.

Research data were collected using the "Structured Description Form", "Modified Pieper Pressure Wound Knowledge Test" and "Satisfaction Scale".

DETAILED DESCRIPTION:
The research was designed in a randomized controlled experimental type in order to determine the effect of mobile application on students' knowledge levels and satisfaction levels about the prevention, treatment and care of pressure injuries.

Research Hypotheses Hypothesis 1 (H1) The knowledge level of nursing students using mobile applications in teaching the care and treatment of pressure injuries is higher than the students receiving education with the classical method.

Hypothesis 2 (H2) Nursing students who receive education using mobile applications in teaching the care and treatment of pressure injuries have higher education satisfaction levels than students who receive education with the classical method.

Universe and Sample The population of the study conducted in the fall semester of the 2020-2021 academic year consisted of students enrolled in the Basic Principles and Practices in Nursing course at a foundation university in Istanbul between March and June 2021 (N=78). Power analysis (NCSS-PASS Statistical package) was performed to determine the number of students who would form the research sample. The sample size was calculated with G power 3.1.9.4, based on similar studies, and it was calculated that at least 28 people should be included in each group, with the pre-acceptance of α error being 5%, research power (power) 80%, and an effect value of 0.77. In this direction, 58 students who met the study criteria formed the sample of the study. In the randomization of the study, students were assigned to the experimental (n=29) and control (n=29) groups according to their numbers in the class list using the www.random.org program. Research data were collected using the "Structured Description Form", "Modified Pieper Pressure Wound Knowledge Test" and "Satisfaction Scale".

ELIGIBILITY:
Inclusion Criteria:

Nursing students;

* be 18 years or older,
* Not having graduated from Health Vocational High School,
* To be registered for the first time in the Basic Principles and Practices in Nursing course, to fully participate in the interventions to be applied in the study.
* Volunteer to participate in the study.

Exclusion Criteria:

Nursing students;

* be under the age of 18,
* Having graduated from Health Vocational High School,
* Having taken the Basic Principles and Practices in Nursing course before,
* Not participating in the initiatives to be implemented in the study,
* Not willing to participate in the study

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
knowledge levels | 2 Months
  Nursing student were informed about the prevention, care and treatment of pressure injuries.
Level of Satisfaction | 2 Month
  Level of Satisfaction: The satisfaction levels of nursing students from the training given about the prevention, care and treatment of pressure injury were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, PhD RN, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Beykent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forehand, J. W., Miller, B., & Carter, H. (2017). Integrating mobile devices into the nursing classroom. Teaching and Learning in Nursing, 12(1), 50-52.
- [Result] Barakat-Johnson, M., Lai, M., Wand, T., & White, K. (2019). A qualitative study of the thoughts and experiences of hospital nurses providing pressure injury prevention and management. Collegian, 26(1), 95-102.
- [Result] Kim SJ, Shin H, Lee J, Kang S, Bartlett R. A smartphone application to educate undergraduate nursing students about providing care for infant airway obstruction. Nurse Educ Today. 2017 Jan;48:145-152. doi: 10.1016/j.nedt.2016.10.006. Epub 2016 Oct 25. PMID 27810633
- [Result] Lee NJ, Chae SM, Kim H, Lee JH, Min HJ, Park DE. Mobile-Based Video Learning Outcomes in Clinical Nursing Skill Education: A Randomized Controlled Trial. Comput Inform Nurs. 2016 Jan;34(1):8-16. doi: 10.1097/CIN.0000000000000183. PMID 26389858